CLINICAL TRIAL: NCT04498130
Title: Designing and Testing the Feasibility of a Theory-Based Intervention to Promote Physical Activity Among Cancer Survivors
Brief Title: Feasibility of a Novel, Theory Based Physical Activity Intervention Among Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21591
Record Dates: First submitted 2020-03-23; First posted 2020-08-04 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cancer Survivors; Exercise; Sedentary Behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-Week Home Exercise Group (Experimental): The 12-week theory-based physical activity intervention will involve mailing participants an exercise manual with health and exercise information (i.e. information about exercising safely, modules related to the social cognitive theory, weekly goal setting worksheets, exercise-tracking logs, etc.), a resistance band, and a standard Omron pedometer. Participants will receive a weekly 30-minute Zoom--based group meetings to discuss different strategies to begin and maintain a consistent exercise routine and access to a social media page to facilitate social support and interaction among the group participants. Participants will be able to join the group if they would like, but it will not be required. Participants will be encouraged to connect with each other to promote social support and social modeling. Lastly participants will receive a weekly exercise video to follow along with on their own time and tailored weekly step goals.
  Interventions: Behavioral: 12-Week Home Exercise Group
- Educational Comparison Group (Active Comparator): The education group participants will receive the same exercise manual, fitness items, exercise videos, and same weekly tailored step goal as the 12-week intervention group. This group will not have weekly zoom discussions, or be a part of the same social media page as the 12-week intervention group. Instead, the education group will be contacted by research staff once a week via telephone to discuss their manuals and activity for the week, and to ensure they have been safely engaging in exercise. A separate social media page will be created for this group, where pre-existing materials related to physical activity recommendations, benefits, other resources, and more will be shared.
  Interventions: Behavioral: Education Comparison Group

INTERVENTIONS:
Behavioral: 12-Week Home Exercise Group — 12 week home-based program consisting of: weekly Zoom group chats; exercise videos; free exercise equipment and pedometer; an exercise manual with worksheets to promote increased physical activity; access to a unique group social media page
  Arms: 12-Week Home Exercise Group
Behavioral: Education Comparison Group — 12 week home-based program consisting of: weekly check-in phone calls; exercise videos; free exercise equipment and pedometer; an exercise manual with worksheets to promote increased physical activity; access to a unique group social media page.
  Arms: Educational Comparison Group

SUMMARY:
As the number of cancer survivors grows and expected survival time increases, the health behaviors of this population are gaining significant attention from the research and public health community. Adoption or maintenance of healthy lifestyles after cancer has the potential to reduce both cancer- and non-cancer-related morbidity and mortality. Exercise adoption and maintenance remains a significant challenge for adults, especially clinical populations such as cancer survivors who may struggle with comorbidities, symptoms and side-effects of the disease or medications, and overall compromised health and functioning. A number of site-based exercise interventions have been conducted to promote physical activity, often using a theoretical basis to design and execute the intervention. Although these programs are successful in exposing cancer survivors to regular physical activity, they often struggle with exercise maintenance after the conclusion of the structured site-based group exercise sessions. The goal of the proposed project is to enhance physical activity engagement among adult cancer survivors by designing a home-based program using the socio-ecological framework and employing constructs from social cognitive theory to guide participants through the project.

ELIGIBILITY:
Inclusion Criteria:

* 30-75 years of age at baseline
* Cancer diagnosis during adulthood (no childhood cancers)
* Low-active (≤ 2 days of 30 minutes of structured exercise/week)
* At least 1 month since last cancer treatment (surgery, chemotherapy and/or radiation)
* No reservations from a doctor/physician/oncologist to engage in physical activity
* Not currently undergoing cancer-related treatment
* No active cancer diagnosis
* Willingness to participate in a 12-week home exercise program
* Willingness to be randomized to either the 12-week home exercise or a 12 week education group
* Access to a laptop/ phone with Zoom web-conferencing software
* An active email address to receive and sign the electronic informed consent
* Willingness to complete study questionnaires before and after the 12-week program, and 3 months after the program
* Fluency in English

Exclusion Criteria:

* Below 30 or above 75 of age at baseline
* Childhood cancer diagnosis only
* High active (> 2 days of 30 minutes of structured exercise/week)
* Cancer treatment within the last month or currently undergoing treatment
* Advised to refrain from physical activity by a doctor/physician/oncologist
* Active cancer diagnosis
* Not willing to participate in a 12-week home exercise group and/or complete study assessments
* Not willing to be randomized into one of the two study groups
* No access to a laptop/phone with Zoom software
* No access to active email
* Not fluent in English

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Zoom-Based Exercise Coaching | 12 weeks
  Participants in the intervention arm will answer Likert-format questions relating to their preference, tolerance and usage of the Zoom-based group meetings to promote physical activity levels. The scale will use a 1-5 rating, with 1 being lowest preference/displeased and 10 being the highest preference/very pleased.
Change in average daily step count | Baseline, 12 weeks, 24 weeks
  Participants will wear a hip-based pedometer for 7 days at baseline, 12 weeks and 24 weeks.
Change in minutes of daily sedentary time | Baseline, 12 weeks, 24 weeks
  The Sedentary Behavior Questionnaire (developed by Rosenberg et al., 2010) will be administered at baseline,12 weeks and 24 weeks to assess participants' time spent sitting. Questions relating to sedentary behavior cover both weekday and weekend sitting time, as well as domain-specific sedentary behaviors (i.e. occupational, transportation, and leisure sitting time).Response options for the amount of time engaged in each behavior include: none, 15 minutes or less, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, or 6 hours or more. For scoring, the time spent in each behavior is converted into hours, and the hours per day for each item are summed separately for weekdays and weekend days. Higher scores indicate higher amounts of daily sitting time.

SECONDARY OUTCOMES:
Use of the exercise manual | 12 weeks
  Participants in both groups will answer Likert-format questions relating to their preference, usage and perceived helpfulness of the study-specific exercise manual. The scale will use a 1-10 rating, with 1 being lowest preference/displeased and 10 being the highest preference/very pleased.
Change in physical activity engagement | Baseline,12 weeks, 24 weeks
  The Godin-Shepard Leisure Time Exercise Questionnaire will be administered at baseline, 12 weeks and 24 weeks to assess individuals' reported weekly frequency of engaging in light, moderate and strenuous vigorous-intensity exercise. For each intensity level, participants will report the number of times per week they engaged in an exercise bout >=10 minutes and the average duration of the bouts. For each intensity level, the number of bouts per week will be multiplied by the average duration per bout to reflect participant's average activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Neha P Gothe, MA, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States